CLINICAL TRIAL: NCT07239609
Title: Acceptance and Commitment Therapy for Individuals With MNCD and Their Care Partners: An In-Person and Telehealth Individual Therapy Approach
Brief Title: ACT for Individuals With MNCD and Their Care Partners
Acronym: ACT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Jonathan Singer, Assistant Professor, Texas Tech University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TexasTechU7
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Depression in Adults; Anxiety Disorder Generalized; Grief
Keywords: Mild Cognitive Impariment; Mild Neurocognitive Disorder; Dyadic intervention
MeSH Terms: conditions — Generalized Anxiety Disorder; Neurocognitive Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance Commitment Therapy (Experimental): Acceptance and Commitment Therapy (ACT) is a form of cognitive-behavioral therapy that aims to enhance psychological flexibility through six core processes: acceptance, cognitive defusion, being present, self-as-context, values clarification, and committed action. Rather than attempting to eliminate difficult thoughts and feelings, ACT encourages individuals to accept them while committing to behavior changes consistent with their personal values.
  Interventions: Behavioral: Acceptance Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance Commitment Therapy — Acceptance and Commitment Therapy (ACT) is a form of cognitive-behavioral therapy that aims to enhance psychological flexibility through six core processes: acceptance, cognitive defusion, being present, self-as-context, values clarification, and committed action. Rather than attempting to eliminate difficult thoughts and feelings, ACT encourages individuals to accept them while committing to behavior changes consistent with their personal values.

SUMMARY:
This project aims to implement and evaluate a dyadic intervention (i.e., acceptance commitment therapy) for persons with AD/ADRD and their care partners. We hypothesize the intervention will be feasible, acceptable, and show preliminary efficacy of the dyadic interveniotns.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) and Alzheimer's Disease Related Dementias (AD/ADRD) are life-limiting, long-term, neurodegenerative conditions estimated to affect more than 6.5 million adults over the age of 65 in the U.S. (Alzheimer's Association, 2023a). A majority of persons with AD/ADRD are over the age of 75 (73%; Alzheimer's Association, 2023a). With an aging population (estimated 1 in 6 people in the world will be over the age of 60 by 2030; World Health Organization, 2022), no known cure, and modern medical advances increasing life expectancy, the prevalence of AD/ADRD continues to rise, an estimated 13.8 million by 2060 (Alzheimer's Association, 2023a). Due to this mostly affecting older adults, 69.1% are living with a comorbid diagnosis (e.g., hypertension; diabetes) (Bennett et al., 2018; Poblador-Plou et al., 2014). AD/ADRD presents a global health crisis, posing profound challenges to not only the individuals with the disease, but has downstream effects on the family unit and the healthcare systems. As number of individuals with AD/ADRD are expected to increase over the next 10 years, it is vital to investigate non-pharmacological interventions for this population in order to improve the negative consequences of this diagnosis. This study aims to bridge this gap by investigating a modified evidence-based intervention, Acceptance Commitment Therapy (ACT), for persons with AD/ADRD and their care partners.

An integral part of an AD/ADRD journey is the care partner, who is usually a spouse or adult child. These care partners provide more than 10 billion hours of care in the United States to individuals with AD/ADRD. This has been found to result in negative outcomes, including high rates of pre-death grief, caregiver burden, and stress. There have been numerous non-pharmacological interventions for these care partners, but few studies have investigated the effects of dyadic interventions for persons with AD/ADRD and their care partners. Dyadic interventions have been found to be effective in improving psychosocial outcomes with persons with other chronic conditions (e.g., cancer) and their care partners (Hu etl a., 2019). The overarching goal of this project is to evaluate if acceptance commitment therapy will have a positive effect on persons recently diagnosed with early stage AD/ADRD.

More specifically, we will:

1. Evaluate the feasibility and acceptability of this shortened ACT program for persons with MCI or MNCD.
2. Assess the preliminary efficacy of this ACT program for persons with MCI or MNCD.
3. Evaluate if this intervention program has positive downstream effects on the care partners.

ELIGIBILITY:
Inclusion Criteria

Inclusion (person with MCI or MNCD):

* 18+
* MMSE= 21-27
* Able to communicate in English

Inclusion (care partner):

* 18+
* Identifies as a care partner of a person with MNCD
* Able to communicate in English
* MMSE= 28-30
* Is a family member or friend of the person with MNCD

Exclusion Criteria

Exclusion (person with MCI or MNCD):

* Currently in an intervention for reducing anxiety or depression related to their dementia
* MMSE= 28+ or less than 21

Exclusion (care partner):

* MMSE= <28
* Is a formal (paid) caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | 6 weeks
  PHQ-9 is used to assess the presence and severity of depressive symptoms.
Geriatric Depression Short From | 6 Weeks
  GDS short is a brief, self-report screening tool designed to identify depressive symptoms in older adults.
The Generalized Anxiety Disorder-7 | 6 weeks
  GAD-7 is used to assess the severity of generalized anxiety symptoms
General Anxiety Scale-10 | 6 Weeks
  The GAS-10 is designed to assess the severity of general anxiety symptoms
Pre-death grief-12 | 6 weeks
  The PG-12 examines pre-death grief for persons with life limiting illnesses and their care partners.

SECONDARY OUTCOMES:
Dyadic Coping Inventory | 6 Weeks
  The DCI assess how couples support each other and cope together with stress.
Short Form Health Survey (SF-12) | 6 Weeks
  The SF-12 measures functional health and well-being
Purpose in Life Scale | 6 Weeks
  The PIL is designed to assess an individual's sense of meaning and purpose in life.
Herth Hope Index | 6 Weeks
  The HHI is designed to measure an individual's level of hope
Inclusion of Other in the Self Scale | 6 Weeks
  The IOS is designed to assess perceived closeness in interpersonal relationships
Perceived Stress Scale | 6 Weeks
  The PSS is a measure the degree to which individuals perceive their lives as stressful
Pittsburgh Sleep Quality Index | 6 Weeks
  The PSQI assess sleep quality and disturbances.
Repeatable Battery for the Assessment of Neuropsychological Status | 6 Weeks
  The RBANS is a neuropsychological assessment designed to evaluate cognitive functioning

IPD SHARING:
Plan to Share IPD: No
The investigators will not be providing any individual participant data. It will all be aggregate